CLINICAL TRIAL: NCT01590017
Title: Feasibility Study of Safety, Toxicity, and Compliance of Concomitant Chemoradiotherapy for HIV-Associated Locally-Advanced Cervical Cancer
Brief Title: Cisplatin and Radiation Therapy in Treating Patients With HIV-Associated Locally Advanced Cervical Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AIDS Malignancy Consortium (Network)
Collaborators: National Cancer Institute (NCI) (NIH); The Emmes Company, LLC (Industry); University of Arkansas (Other); Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMC-081; CDR0000732629 (Other: NCI); UM1CA121947 (NIH)
Record Dates: First submitted 2012-05-01; First posted 2012-05-02 (Estimated); Results first posted 2019-08-07 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2019-07

CONDITIONS: Cervical Cancer; Acquired Immunodeficiency Syndrome
Keywords: stage IB cervical cancer; stage IIA cervical cancer; stage IIB cervical cancer; stage III cervical cancer; stage IVA cervical cancer; cervical adenocarcinoma; cervical adenosquamous cell carcinoma; cervical squamous cell carcinoma; HIV infection
MeSH Terms: conditions — Uterine Cervical Neoplasms; Acquired Immunodeficiency Syndrome; HIV Infections | interventions — Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cistplatin and Radiation Therapy (Experimental): Cisplatin 40 mg/m2 (max = 70 mg) IV over 30-60 minutes given weekly on days 1, 8, 15, 22, 29 and 36 for a total of 6 weekly cycles. Radiation therapy over 8 weeks: External pelvic radiation therapy (41.4-45.0 Gy/1.8 Gy per fraction/23-25 fractions/five weeks), intracavitary brachytherapy (low dose: 35-43.6 Gy/1-2 implants; high dose: 18-28 Gy/2-4 implants), with parametrial boost to involved parametria (5.40 - 9.00 Gy/1.8 Gy/3-5 fractions/3-5 days).
  Interventions: Drug: cisplatin; Radiation: external beam radiation therapy

INTERVENTIONS:
Drug: cisplatin
Radiation: external beam radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x rays to kill tumor cells. Giving cisplatin together with radiation therapy may be an effective treatment for cervical cancer.

PURPOSE: This trial studies how well cisplatin and radiation therapy work in treating participants with HIV-associated locally advanced cervical cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine if it is feasible to administer a regimen of cisplatin/radiotherapy in HIV-infected women with locally advanced cervical cancer (LACC) on antiretroviral therapy (ART).
* To evaluate the safety and tolerability of concomitant chemoradiotherapy with cisplatin in HIV-infected women with LACC who are also receiving concomitant ART.

Secondary

* To determine the 1-year progression-free survival (PFS) of HIV-infected women with LACC Stage IB, II, III, or IVA who receive weekly cisplatin concomitant with radiotherapy and ART. (Exploratory)
* To describe the quality of life (QOL) of enrolled participants via assessments before, immediately after, and at 3 and 9 months after completion of therapy, using QOL metrics that have been validated in similar populations. (Exploratory)
* To describe the effects of treatment on participants' CD4 counts, HIV viral load, and concurrent AIDS-defining conditions. (Exploratory)
* To describe cervical cancer recurrence patterns in HIV-infected participants with LACC defined as loco-regional and/or distant recurrences. (Exploratory)
* To determine 1-year overall survival and causes of death (i.e., cancer-related, HIV-related, or other). (Exploratory)
* To collect serum, cytology, and tissue for future studies specific to cervical and anal disease. (Exploratory)
* To evaluate the effects of weekly cisplatin concomitant with radiotherapy on adherence to ART. (Exploratory)

OUTLINE: This is a multicenter study.

Participants receive cisplatin IV over 30-60 minutes on days 1, 8, 15, 22, 29, and 36 (6 weeks total). Participants also undergo whole pelvic radiotherapy (WPRT) 5 days a week for 5 weeks followed by intracavitary brachytherapy.

Participants complete the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ)-30 and the Cervical Cancer Module (QLQ-CX24) at baseline and periodically during study treatment.

After completion of study treatment, participants are followed up every 3 months for 12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Participants (who have been adequately clinically staged by standard clinical guidelines) with primary, untreated, histologically confirmed, documented invasive squamous cell carcinoma, adenocarcinoma, or adenosquamous carcinoma of the uterine cervix, stages IB2, IIA, IIB, IIIA, IIIB, and IVA (Stage IIA tumors must be greater than 4 cm)
* HIV-1 infection, documented by any licensed rapid HIV test or HIV enzyme or chemiluminescence immunoassay (E/CIA) test kit at any time prior to study entry and confirmed by a licensed western blot or a second antibody test by a method other than the initial rapid HIV and/or E/CIA, or by HIV-1 antigen, plasma HIV-1 ribonucleic acid (RNA) viral load

  * NOTE: the term "licensed" refers to a United States (U.S) Food and Drug Administration (FDA)-approved kit or for sites located in countries other than the United States, a kit that has been certified or licensed by an oversight body within that country and validated internally
  * WHO (World Health Organization) and CDC (Centers for Disease Control and Prevention) guidelines mandate that confirmation of the initial test result must use a test that is different from the one used for the initial assessment; a reactive initial rapid test should be confirmed by either another type of rapid assay or an E/CIA that is based on a different antigen preparation and/or different test principle (e.g., indirect versus competitive), or a western blot or a plasma HIV-1 RNA viral load
* No participants with carcinoma of the cervical stump

PATIENT CHARACTERISTICS:

* Hemoglobin ≥ 10 g/dL (6.2 mmol/L)
* Platelet count ≥ 100,000/mm³ (100 x 10^9/L)
* Absolute neutrophil count (ANC) ≥ 1000/mm³ (1.0 x 10^9/L) (participants receiving transfusion, erythropoietin, or myeloid growth factor support will be eligible for this study)
* Creatinine clearance ≥ 60 mL/min (1.00 mL/s) calculated by the Cockcroft-Gault equation for women
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 times upper limit of normal (ULN)
* Total bilirubin ≤ 2 times ULN unless related to antiretroviral use (e.g., atazanavir and indinavir), then the direct bilirubin must be ≤ 2 times ULN
* Ability to understand and the willingness to provide informed consent to participate
* Karnofsky performance status of ≥ 60%
* Participants of childbearing potential, defined as a sexually mature woman who has not undergone a hysterectomy or bilateral oophorectomy or has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months), must have a negative urine or serum pregnancy test within 3 weeks prior to enrollment and agree to use an effective form of contraception (e.g., barrier contraception, highly effective hormonal contraception)
* Life expectancy of greater than 12 months
* No acute active (such as tuberculosis or malaria), serious, uncontrolled infection; participants with a CD4 count < 50/mm³ (0.05 x 10^9/L) will be excluded if they have had an opportunistic infection within the past 3 months, or if there is evidence of resistance to antiretroviral therapy (i.e., HIV viral load ≥ 400 copies/mL despite combination antiretroviral therapy for at least 4 months)
* No prior invasive malignancy other than LACC diagnosed within the past 24 months, excluding anal intraepithelial neoplasia, non-melanoma skin carcinoma, or Kaposi sarcoma that has not required systemic chemotherapy within the past 24 months
* No pregnancy or breast-feeding
* No medical or psychiatric illness that precludes ability to give informed consent or is likely to interfere with the ability to comply with the protocol stipulations
* No participants with circumstances that will not permit completion of the study or required follow-up; for instance, if travel to and from treatment site is an issue
* No participants with cardiovascular disease manifested as:

  * History of myocardial infarction
  * Unstable angina
  * Currently taking medication for treatment of angina
  * History of coronary artery bypass surgery
  * New York Heart Association class 3 or 4 heart failure

PRIOR CONCURRENT THERAPY:

* See Patient Characteristics
* All patients must be prescribed combination antiretroviral therapy with the goal of virological suppression using an acceptable regimen that adheres to national guidelines for treatment of HIV infection

  * Non-suppressed, treatment-experienced patients, defined as patients with a viral load > 400 copies/mL who have been on antiretroviral therapy for more than 4 months, can be enrolled if a genotype assay is performed and an acceptable regimen is prescribed based on the genotyping results
* Patients who undergo emergency radiation therapy prior to enrollment may participate at the investigator's discretion
* No participants who have undergone hysterectomy
* No concurrent intensity-modulated radiotherapy or interstitial brachytherapy

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2014-04-01 (Actual); Primary Completion 2017-04-20 (Actual); Study Completion 2017-04-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark H. Einstein, MD, MS, Principal Investigator — Albert Einstein College of Medicine
Locations (2):
- Clinical HIV Research Unit, a Division of the Wits Health Consortium (Pty) Ltd, Johannesburg, South Africa
- University of Zimbabwe Clinical Research Centre / Parirenyatwa Hospital, Harare, Zimbabwe

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cistplatin and Radiation Therapy: Cisplatin 40 mg/m2 (max = 70 mg) IV over 30-60 minutes given weekly on days 1, 8, 15, 22, 29 and 36 for a total of 6 weekly cycles. Radiation therapy over 8 weeks: External pelvic radiation therapy (41.4-45.0 Gy/1.8 Gy per fraction/23-25 fractions/five weeks), intracavitary brachytherapy (low dose: 35-43.6 Gy/1-2 implants; high dose: 18-28 Gy/2-4 implants), with parametrial boost to involved parametria (5.40 - 9.00 Gy/1.8 Gy/3-5 fractions/3-5 days).
  cisplatin
  external beam radiation therapy
Period: Overall Study
Arm/Group | Cistplatin and Radiation Therapy
Started | 41
Completed | 37
Not Completed | 4
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1
Not completed — Lack of Efficacy | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Population: Patients who enrolled in the study
Arm/Group | Cistplatin and Radiation Therapy
Number analyzed (Participants) | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.2 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 41
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  South Africa | 15
  Zimbabwe | 26

OUTCOME MEASURES:

1. Primary Outcome: Treatment Completion Rate
Description: Number of participants who completed therapy
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Cistplatin and Radiation Therapy
Number analyzed (Participants) | 41
Participants | 37

2. Primary Outcome: Patients With Adverse Events
Description: Number of patients who experienced one or more adverse events
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cistplatin and Radiation Therapy
Number analyzed (Participants) | 41
Participants | 39

ADVERSE EVENTS:
Time Frame: One year
Arm/Group | Cistplatin and Radiation Therapy
All-Cause Mortality (participants affected / at risk) | 7/41
Serious Adverse Events (participants affected / at risk) | 10/41
Other Adverse Events (participants affected / at risk) | 39/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cistplatin and Radiation Therapy (N=41)
Vomiting (Gastrointestinal disorders) | 2
Metastatic Cancer of the uterine cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5
Thromboembolic event (Vascular disorders) | 2
anemia (Blood and lymphatic system disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Death NOS (General disorders) | 1
Flu-like symptoms (General disorders) | 1
Neutrophil count decreased (Investigations) | 1
Chronic kidney disease (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cistplatin and Radiation Therapy (N=41)
Anemia (Blood and lymphatic system disorders) | 13
Constipation (Gastrointestinal disorders) | 4
Diarrhea (Gastrointestinal disorders) | 5
Hemorrhoids (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 3
Infections (Infections and infestations) | 4
Urinary tract infection (Infections and infestations) | 3
Lymphocyte decreased (Investigations) | 15
Neutrophil count decrease (Investigations) | 36
Platelet count decreased (Investigations) | 17
White blood cell decreased (Investigations) | 15
Weight loss (Investigations) | 8
Hypokalemia (Metabolism and nutrition disorders) | 3
Hypomagnesia (Metabolism and nutrition disorders) | 7
Hyponatremia (Metabolism and nutrition disorders) | 11
Pain (Musculoskeletal and connective tissue disorders) | 3
Metastatic cervix cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Chronic kidney disease (Renal and urinary disorders) | 3
Urinary tract pain (Renal and urinary disorders) | 6
Vaginal discharge (Reproductive system and breast disorders) | 7
Vaginal hemorrhage (Reproductive system and breast disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Desquamation of the perineum (Skin and subcutaneous tissue disorders) | 3
Hypertension (Vascular disorders) | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-02-20): https://cdn.clinicaltrials.gov/large-docs/17/NCT01590017/Prot_SAP_000.pdf